CLINICAL TRIAL: NCT00002774
Title: Randomized Phase 2 Trial of Tirapazamine and the Role of Tumor Hypoxia in Advanced Squamous Head and Neck Cancer
Brief Title: Radiation Therapy and Combination Chemotherapy in Treating Patients With Stage III or Stage IV Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: IRB-12503; CA67166 (Other Grant/Funding Number: Public Health Service / National Cancer Institute); NCI-T94-0119O (Other: National Cancer Institute); CDR0000064752; SQL 72951 (Other: Stanford IRB legacy identifier)
Record Dates: First submitted 2000-04-06; First posted 2004-04-06 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Squamous Neck Carcinoma of the Head and Neck Cancer (SCCHN)
Keywords: stage III; stage IV; recurrent
MeSH Terms: conditions — Head and Neck Neoplasms; Recurrence | interventions — Tirapazamine; Cisplatin; Fluorouracil; Radiotherapy

ARMS (2):
- Tirapazamine + cisplatin + 5-FU (Experimental): 2 cycles of induction chemotherapy (tirapazamine, cisplatin, and 5-fluorouracil [5-FU]) followed by simultaneous chemoradiotherapy (tirapazamine, cisplatin, and 5-FU)
  Interventions: Drug: Tirapazamine; Drug: Cisplatin; Drug: 5-fluorouracil; Radiation: Radiotherapy (RT)
- Cisplatin + 5-FU (Active Comparator): 2 cycles of induction chemotherapy (cisplatin + 5-fluorouracil [5-FU]) followed by simultaneous chemoradiotherapy (cisplatin + 5-FU)
  Interventions: Drug: Cisplatin; Drug: 5-fluorouracil; Radiation: Radiotherapy (RT)

INTERVENTIONS:
Drug: Tirapazamine — Tirapazamine is a benzotriazine with selective cytotoxicity for hypoxic cells. Under hypoxic conditions, it undergoes a 1-electron reduction to form a cytotoxic free radical that poisons topoisomerase II and causes DNA breaks, chromosomal aberrations, and cell death.
  Tirapazamine was administered on Days 1 and 22 prior to the administration of neoadjuvant cisplatin and on Days 43, 45, 47, 71, 73, and 75 within 1 or 2 hours prior to each simultaneous cisplatin dose.
  Tirapazamine dose was as follows:
  Level 1 - 300 mg/m2 during the induction phase and 160 mg/m2 during the simultaneous phase (n = 4)
  Level 2 - 330 mg/m2 during the induction phase and 260 mg/m2 during the simultaneous phase (n = 4)
  Level 3 - 300 mg/m2 during the induction phase and 220 mg/m2 during the simultaneous phase (n = 25)
  Other Names: Tirazone; TPZ; SR 4233; 3-amino-1,4-benzotriazine-1-N-oxide; WIN 59074
  Arms: Tirapazamine + cisplatin + 5-FU
Drug: Cisplatin — The simultaneous chemoradiotherapy (CRT) regimen included cisplatin 20 mg/m2 administered 3 times per week.
  Other Names: Cisplatinum; Cis-diamminedichloroplatinum(II); CDDP
Drug: 5-fluorouracil — 100 mg/m2 per day on Days 1 and 22, and continuous infusion (CI) 5-FU at a dose of 1000 mg/m2 per day for 120 hours per cycle starting on Days 1 and 22.
  The simultaneous chemoradiotherapy (CRT) regimen included continuous infusion (CI) 5-FU 600 mg/m2 per day for 96 hours per cycle in Weeks 1 and 5 of RT.
  Other Names: 5-FU
Radiation: Radiotherapy (RT) — During the CRT regimen, RT was given within 3 hrs of the tirapazamine infusion. The dose for the parallel opposed fields was 2 Gy/fraction/day given 5 dys/week up to a total dose of 66-70 Gy at the target lesion. The dose to the supraclavicular region was 50 Gy at a depth of 3 cm, delivered in 25 fractions. Supervoltage photons (≥4 megavolts) were used to treat both locations.
  After 50 Gy were delivered to the primary site and regional lymph nodes, all sites were reassessed for clinical response by physical exam, direct fiber optic evaluation, and radiographic imaging (CT or MRI).
  Subjects with a CR at both the primary site and the neck completed RT treatment to a total dose ≥66 Gy to the primary site and the involved lymph node(s). Subjects with a CR at the primary site but a partial response (PR) at the neck completed RT treatment to the primary site followed by neck dissection. Subjects with a PR at the primary site stopped radiation at 50 Gy and underwent salvage surgery.

SUMMARY:
PURPOSE: Randomized phase 2 trial to compare the effectiveness of chemo-radiation therapy (RT + cisplatin + 5-FU) with or without tirapazamine for the treatment of patients with stage III or IV squamous cell carcinomas of the head and neck cancer (SCCHN).

RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. Radiation therapy uses high-energy x-rays to damage tumor cells.

Tirapazamine may increase the effectiveness of chemotherapy and radiation therapy by making tumor cells more sensitive to therapy.

DETAILED DESCRIPTION:
Subjects were stratified according to pO2 values (high vs low), and randomized to 1 of 2 treatment arms, differing by the addition of tirapazamine to the therapeutic regimen. Treatment consists of two 21-day cycles of induction chemotherapy, followed by radiotherapy (RT).

Induction chemotherapy was cisplatin 100 mg/m2 per day administered over 4 hours on Study Days 1 and 22 (ie, 1st day of both induction cycles) with continuous infusion (CI) 5-FU at a dose of 1000 mg/m2 per day for 120 hours per cycle starting on Study Days 1 and 22 (ie, days 1 to 5 of both induction cycles).

Patients who achieve at least partial response proceeded to chemoradiotherapy (CRT) consisting of localized RT + cisplatin IV + 5-FU +/- tirapazamine. Location of RT was based on whether the site had a CR or PR. Radiotherapy began on day 43 (week 1), and continued for 5.5 weeks. Subjects with no response or progressive disease proceeded to salvage surgery.

A total of 63 patients were accrued for this study over approximately 5 years. 1 subject withdrew consent prior to treatment for personal reasons.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Biopsy proven squamous cell carcinoma of the following head and neck sites:

Hypopharynx Oral cavity Larynx Oropharynx Nasal cavity Unknown primary Paranasal sinus

Histologically proven poorly-differentiated carcinoma of the following head and neck sites:

Hypopharynx Oral cavity Larynx Oropharynx Nasal cavity Paranasal sinus Stage III/IV (T0-4 N1-3 M0-2) disease

PATIENT CHARACTERISTICS:

WBC at least 3,000/mm3 Bilirubin no greater than 2.0 mg/dL AST no greater than 100 U/L Creatinine no greater than 2.0 mg/dL Creatinine clearance at least 60 mL/min (patients in Group N2-N3) No second malignancy within 5 years except curatively treated nonmelanomatous skin carcinoma No prior RT or chemotherapy, except prior radiotherapy to primary tumor allowed Not pregnant or nursing. Negative pregnancy test required Effective contraception required of fertile women Subjects with unknown primary cancers who had metastatic cervical lymph nodes are eligible Signed informed consent previously approved by the Institutional Review Board.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 1996-06; Primary Completion 2000-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Complete response rate (CRR) | 12 weeks
  Compare the CRR following CRT with or without tirapazamine in patients with squamous cell carcinoma of the head and neck.

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
  Survival was assessed at 5 years post-treatment.
Cause-specific survival (CSS) | 5 years
  CSS is also known as disease-specific survival (DSS), and in this study represents cancer survival from diagnosis until death due to cancer, in the absence of other causes of death. All other causes of death are censored.
Rate of freedom from recurrence (FFR) | 5 years
  FFR is the period until first treatment failure, and typically includes failure to achieve CR, but does not include deaths.

CONTACTS AND LOCATIONS:
Overall Officials: Harlan A. Pinto, MD, Study Chair — Stanford University
Locations (2):
- United States (2):
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford University Medical Center, Stanford, California

REFERENCES:
- [Result] Le QT, Taira A, Budenz S, Jo Dorie M, Goffinet DR, Fee WE, Goode R, Bloch D, Koong A, Martin Brown J, Pinto HA. Mature results from a randomized Phase II trial of cisplatin plus 5-fluorouracil and radiotherapy with or without tirapazamine in patients with resectable Stage IV head and neck squamous cell carcinomas. Cancer. 2006 May 1;106(9):1940-9. doi: 10.1002/cncr.21785. PMID 16532436